CLINICAL TRIAL: NCT04051671
Title: Effects of Dual-transcranial Direct Current Stimulation During Physical Therapy in Sub-acute Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: National Research Council of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MU-CIRB 2019/045.1102
Record Dates: First submitted 2019-08-08; First posted 2019-08-09 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS & PT (Experimental): Dual transcranial direct current stimulation (tDCS) will be applied over the leg motor area (M1) during the first 20 mins of conventional physical therapy (about 1 hours). Anodal on affected hemisphere, Cathodal on unaffected hemisphere. Current intensity is fixed at 2 mA and current will flow continuously during 20. Physical therapist will give an intervention program exactly the same in all cases. The scope of intervention is administered to improve strength of weakened and postural lower limbs muscles such as trunk muscles, hip flexors/extensors/abductors, knee flexors/extensors.
  Interventions: Device: Transcranial direct current stimulation
- Sham tDCS & PT (Active Comparator): Dual transcranial direct current stimulation (tDCS) will be applied over the leg motor area (M1) during the first 20 mins (sham mode) of conventional physical therapy (about 1 hours). Anodal on affected hemisphere, Cathodal on unaffected hemisphere. Physical therapist will give an intervention program exactly the same in all cases. The scope of intervention is administered to improve strength of weakened and postural lower limbs muscles such as trunk muscles, hip flexors/extensors/abductors, knee flexors/extensors.
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — Dual Active/sham tDCS will be applied over the leg motor area (M1) during the first 20 mins of conventional physical therapy. Anodal on affected hemisphere, Cathodal on unaffected hemisphere. Each participant will complete two experiments (active/sham tDCS). The interval between two experiments is at least 2 weeks. The two experiments will be performed in random order for each subject.

SUMMARY:
The aim of the present study is to evaluate the possible effect of using dual-tDCS applied during conventional physical therapy on lower limb function in stroke patients.

DETAILED DESCRIPTION:
Recently dual-tDCS applied before the conventional physical therapy show positive effect of lower limb performance. However to explore the time during which dual-tDCS can be combined with physical therapy to maximize motor performance is required. Results from the present study with be compared with our previous study that used dual-tDCS applied before physical therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age range 18-75 years.
2. First ever-ischemic lesion in the territory of middle cerebral artery or anterior cerebral artery. CT scan/MRI result is thus required.
3. Sub acute phase of stroke (less than 6 months)
4. Able to sit-to-stand and stand-to-sit independently
5. Able to walk without physical assistance at least 6 m
6. Free of any neurological antecedent, unstable medical conditions or condition that may increase the risk of stimulation such as epilepsy

Exclusion Criteria:

1. Pre-stroke disability
2. Pregnant
3. Be unable to understand the instruction
4. No clear neurological antecedent history or psychiatric disorder
5. Excessive pain in any joint of the paretic limb (numerical pain rating score > 7)
6. Presence of intracranial metal implantation, cochlea implant, or cardiac pacemaker
7. Subjects are participating in the other protocol or receiving alternative treatment such as acupuncture

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2019-10-06 (Actual); Study Completion 2019-11-06 (Actual)

PRIMARY OUTCOMES:
Five-Times-Sit-To-Stand test (FTSST) | 5 minutes
  sling. Subjects will be instructed as the following "I want you to stand up and sit down 5 times as quickly as you can when I say 'Go'." Subjects must be fully standing between repetitions. Timing will begin at "GO" and ends when the patient's buttocks touch the seat after the fifth sit-to-stand.
Timed Up & Go test (TUG) | 5 minutes
  Subjects will sits on the chair and place their back against the chair. Timing will begin at "GO", the subjects will be asked to walk 3m, turn, walk back, and sit down. The stopwatch stops when the patient's buttocks touch the seat.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty ofPhysical Therapy, Mahidol University, Salaya, Nakonpathom, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Klomjai W, Aneksan B. A randomized sham-controlled trial on the effects of dual-tDCS "during" physical therapy on lower limb performance in sub-acute stroke and a comparison to the previous study using a "before" stimulation protocol. BMC Sports Sci Med Rehabil. 2022 Apr 15;14(1):68. doi: 10.1186/s13102-022-00463-9. PMID 35428346